CLINICAL TRIAL: NCT00455806
Title: Randomized, Controlled, Multicenter Phase III Study for the Efficacy and Tolerability of Triple Therapy With Esomeprazole, Moxifloxacin and Amoxicillin for Rescue Therapy of Helicobacter Pylori Infection
Brief Title: Esomeprazole, Moxifloxacin and Amoxicilin for Rescue Therapy of Helicobacter Pylori Infection
Acronym: ESAMOX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESAMOX_01_2007; EudraCT Numberr 2006-004323-10
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-03

CONDITIONS: Helicobacter Pylori Infection; Chronic Gastritis
Keywords: Helicobacter pylori; rescue therapy; eradication therapy; esomeprazole; moxifloxacin; resistance
MeSH Terms: interventions — Esomeprazole; Moxifloxacin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: esomeprazole
Drug: moxifloxacin
Drug: amoxicillin

SUMMARY:
Successful H. pylori eradication therapy remains a challenge in medical practice. Despite promising data for first-line, second-line and rescue treatment options based on clinical trials as well as guidelines and expert recommendations, success rates can often not be reproduced in general practice. Rescue options for patients with failed initial or second-line therapy are definitely needed. The new fluoroquinolone moxifloxacin may represent an effective and save treatment option (in combination with a PPI and amoxicillin) for rescue therapy of H- pylori positive patients.However, optimal duration of therapy (7-day course vs 14-day course) has to be determined

DETAILED DESCRIPTION:
Successful H. pylori eradication therapy remains a challenge in medical practice. Currently, a PPI - based triple therapy containing clarithromycin, amoxicillin or nitroimidazole given for 7 days is the recommended first line treatment approach with an expected eradication success rate of approximately 80%. As second-line treatment option in case of failure, a RBC-based quadruple therapy is currently recommended curing another 80% of patients, leaving a subset of patients with persistent H. pylori infection. Resistance to fluoroquinolones is low in most countries,hence these compounds are potential candidates for second-line and rescue treatment. The new fluoroquinolone moxifloxacin launched by Bayer in 1999 for the treatment of respiratory tract infections, has a broad antibacterial spectrum comparable to levofloxacin but fewer phototoxic and central nervous system excitatory effects. The possible role of moxifloxacin in H. pylori eradication is since under clinical investigation

ELIGIBILITY:
Inclusion Criteria:

* male/female, age >/=18 years
* Helicobacter pylori infection proven by histology and culture
* indication for eradication therapy according to the Maastricht-III
* at least one failed prior eradication attempt
* pretherapeutic resistance testing (culture)
* written informed consent

Exclusion Criteria:

* in vitro resistance to moxifloxacin or amoxicillin
* current complicated peptic ulcer disease
* daily intake of NSAIDs
* co-medication with drugs known to interact with the study medication
* history of gastric surgery/vagotomy
* medical treatment for depression, known suicide attempt
* severe cardiological diseases such as bradyarrythmia, QT changes
* malignant disease
* gravidity, nursing
* women with child bearing potential must perform contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2007-01; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a combination of esomeprazole (E), moxifloxacin (M) and amoxicillin (A) for third line therapy of H. pylori infection.
Comparison of EMA 7 days versus EMA 14 days. Hypothesis: superiority of EMA 14 days 4 weeks after end of eradication therapy

SECONDARY OUTCOMES:
Tolerability,safety, post treatment resistance, influence of host genetics (CYP status) and pathogenicity factors of H. pylori on treatment success.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Miehlke, MD, PhD, Principal Investigator — Medical Department I, Gastroenterology, Universityhospital, Technical University Dresden; Norbert Lehn, MD, PhD, Study Chair — Institue for Medical Microbiology, University of Regensburg; Enno Jacobs, MD, PhD, Study Chair — Institute for Medical Microbiology, Technical University of Dresden; Manfred Stolte, MD, PhD, Study Chair — Institute for Pathology, Klinikum Bayreuth
Locations (9):
- Germany (9):
  - Gastroenterologist, private praxis, Cologne
  - Med. Dept. I, Gastroenterology, University Hospital, Technical University of Dresden, Dresden
  - Gastroenterologist / private praxis, Görlitz
  - Medical Department, University Homburg/Saar, Homburg/Saar
  - Medical Dept. I, University Hpspital Kiel, Kiel
  - Gastroenterologist / private praxis, Munich
  - Technical University of Munich, Medical Dept. II, Munich
  - Gastroenterologist / private praxis, Oldenburg
  - Med. Department, Jung-Stilling Krankenhaus, Siegen

REFERENCES:
- [Background] Morgner A, Labenz J, Miehlke S. Effective regimens for the treatment of Helicobacter pylori infection. Expert Opin Investig Drugs. 2006 Sep;15(9):995-1016. doi: 10.1517/13543784.15.9.995. PMID 16916269
- [Background] Miehlke S, Hansky K, Schneider-Brachert W, Kirsch C, Morgner A, Madisch A, Kuhlisch E, Bastlein E, Jacobs E, Bayerdorffer E, Lehn N, Stolte M. Randomized trial of rifabutin-based triple therapy and high-dose dual therapy for rescue treatment of Helicobacter pylori resistant to both metronidazole and clarithromycin. Aliment Pharmacol Ther. 2006 Jul 15;24(2):395-403. doi: 10.1111/j.1365-2036.2006.02993.x. PMID 16842467
- [Background] Miehlke S, Schneider-Brachert W, Bastlein E, Ebert S, Kirsch C, Haferland C, Buchner M, Neumeyer M, Vieth M, Stolte M, Lehn N, Bayerdorffer E. Esomeprazole-based one-week triple therapy with clarithromycin and metronidazole is effective in eradicating Helicobacter pylori in the absence of antimicrobial resistance. Aliment Pharmacol Ther. 2003 Oct 15;18(8):799-804. doi: 10.1046/j.1365-2036.2003.01764.x. PMID 14535873
- [Background] Miehlke S, Bayerdorffer E, Graham DY. Treatment of Helicobacter pylori infection. Semin Gastrointest Dis. 2001 Jul;12(3):167-79. PMID 11478749
- [Background] Cheon JH, Kim N, Lee DH, Kim JM, Kim JS, Jung HC, Song IS. Efficacy of moxifloxacin-based triple therapy as second-line treatment for Helicobacter pylori infection. Helicobacter. 2006 Feb;11(1):46-51. doi: 10.1111/j.0083-8703.2006.00371.x. PMID 16423089
- [Background] Nista EC, Candelli M, Zocco MA, Cazzato IA, Cremonini F, Ojetti V, Santoro M, Finizio R, Pignataro G, Cammarota G, Gasbarrini G, Gasbarrini A. Moxifloxacin-based strategies for first-line treatment of Helicobacter pylori infection. Aliment Pharmacol Ther. 2005 May 15;21(10):1241-7. doi: 10.1111/j.1365-2036.2005.02412.x. PMID 15882245
- [Background] Di Caro S, Ojetti V, Zocco MA, Cremonini F, Bartolozzi F, Candelli M, Lupascu A, Nista EC, Cammarota G, Gasbarrini A. Mono, dual and triple moxifloxacin-based therapies for Helicobacter pylori eradication. Aliment Pharmacol Ther. 2002 Mar;16(3):527-32. doi: 10.1046/j.1365-2036.2002.01165.x. PMID 11876707
- [Background] Megraud F, Lamouliatte H. Review article: the treatment of refractory Helicobacter pylori infection. Aliment Pharmacol Ther. 2003 Jun 1;17(11):1333-43. doi: 10.1046/j.1365-2036.2003.01592.x. PMID 12786627